CLINICAL TRIAL: NCT01700296
Title: COPD, Inflammation and Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mimi Christiansen, Medical Doctor, Naestved Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 34431
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): "Standard Care": finishing treatment for AECOPD in hospital and after hospital discharge to further control by the GP. In case of severe symptoms and / or airway obstruction (measured by FEV1) refer patients for follow-up in lung clinic. The subjects are recorded with the same subjective, clinical, paraclinical and invasive parameters as the "Best care" group
- Best care (Experimental): "Best Care": subjects are randomly assigned to the "Best care" regardless MRC class and severity of symptoms through:
  1. 10 weeks of rehabilitation (2 hours, 2 times a week) by Region Zealand's instructions on sundhed.dk. COPD rehabilitation includes physical exercise, smoking cessation, medication, nutrition education and psychosocial support and patient education. Rehabilitation provided by a multidisciplinary effort with lung nurse, dietician and physiotherapist according to national and international guidelines (1.5) (6) (24) (25)
  2. Outpatient follow-up every 3 months, a total of 5 visits, and during these visits various subjective, clinical, paraclinical and invasive parameters.
  Interventions: Behavioral: Best care

INTERVENTIONS:
Behavioral: Best care — "Best Care": subjects are randomly assigned to the "Best care" regardless MRC class and severity of symptoms through:
  1. 10 weeks of rehabilitation (2 hours, 2 times a week) by Region Zealand's instructions on sundhed.dk. COPD rehabilitation includes physical exercise, smoking cessation, medication, nutrition education and psychosocial support and patient education. Rehabilitation provided by a multidisciplinary effort with lung nurse, dietician and physiotherapist according to national and international guidelines (1.5) (6) (24) (25)
  2. Outpatient follow-up every 3 months, a total of 5 visits, and during these visits various subjective, clinical, paraclinical and invasive parameters.
  Arms: Best care

SUMMARY:
Patients with chronic obstructive pulmonary disease, also known as COPD or emphysema, is like any other with a chronic illness not only affected by the physical discomfort the illness gives. For COPD patients that is: accelerated loss of lung function, conditioning and increased mortality: 25% of patients hospitalized with COPD exacerbation die 12 months later.

Patients are also characterized by various psychological factors such as reduced quality of life, depression, etc.

Therefore, everywhere in the country newly diagnosed COPD patients are offered rehabilitation in Region Zealand which consists of 10 weeks of classes 2 hours, 2 times a week with physical exercise, smoking cessation, medication, nutrition education and psychosocial support and patient education based on the National Health Service and international recommendations.

In the literature, the effect of rehabilitation on quality of life was measured using a questionnaire (St. George Respiratory Questionnaire (SGRQ)), and the increase in function has been measured using a walk test, but there are no studies which look at the effect on inflammation lungs.

It is important for COPD patients is to prevent exacerbations of the disease, which sometimes requires hospitalization and sometimes treated by their own doctor. It has been proven that inflammation in the lungs is associated with disease severity and exacerbation frequency, and therefore we would like to investigate whether both rehabilitation, close monitoring of patients with time in the pulmonary clinic every 3 months, and instruction in self-administration of medication (antibiotics and corticosteroids) have an effect on especially inflammation in the lungs, number of exacerbations, mortality, lung function and walking capacity.

ELIGIBILITY:
Inclusion Criteria:

* The study includes consecutive patients over 18 years admitted to the Medical dept, Næstved hospital with AECOPD (2 of 3 symptoms: increased breathlessness, sputum or purulens thereof) on the basis of known COPD (post-bronchodilator FEV1 <80% and FEV1/FVC <70% ; measured in stable phase, ie. earlier than 4 weeks after AECOPD). Patients included during hospitalization for AECOPD

Exclusion Criteria:

* Patients can not participate if they have asthma (post-bronchodilator FEV1 increased by> 15%), are pregnant, nursing, has known serious comorbidities (eg cancer, chronic liver cirrhosis or hepatitis) or cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
IL-8 in Sputum | 1 year

SECONDARY OUTCOMES:
IL-8 in serum IL-8 in the BAL fluid | 1 year

OTHER OUTCOMES:
walking distance | 1 year
exacerbation frequency | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Naestved Sygehus, Næstved, Denmark